CLINICAL TRIAL: NCT00684684
Title: A Safety and Feasibility Study of the Chartis System During Diagnostic Bronchoscopy
Brief Title: Safety and Feasibility Study of the Chartis System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmonx Corporation (Industry)
Responsible Party: Carol Anne Yarbrough, RN, Director, Clinical Affairs, Pulmonx, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRT01028
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Bronchoscopy
Keywords: Bronchoscopy; Clinically indicated for routine diagnostic bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Chartis System

INTERVENTIONS:
Device: Chartis System — Assessment of airway flow and pressure

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of the Chartis System in measuring air flow and pressures in isolated lung compartments during bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo clinically indicated routine diagnostic bronchoscopy

Exclusion Criteria:

* Hyperexcretive chronic bronchitis or excessive sputum secretion
* Active pulmonary infection
* FEV1 <20% predicted
* FVC <50% predicted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Adverse events | Until discharge or 24 hours post procedure

SECONDARY OUTCOMES:
Technical success | During procedure

CONTACTS AND LOCATIONS:
Overall Officials: Felix Herth, MD, Principal Investigator — Thoraxklinik am Universitatsklinikum Heidelberg
Locations (1):
- Thoraxklinik am Universitatsklinikum Heidelberg, Heidelberg, Germany